CLINICAL TRIAL: NCT00456560
Title: A Phase I, Randomized, Two-Period, Single-Center Study to Assess the Effect of CYP2D6 and CYP2C19 Inhibitors on a Single Oral Dose of AV650 (300 mg) in Healthy Subjects
Brief Title: AV650 Drug-Drug Interaction Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Avigen (Industry)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: AV650-019
Record Dates: First submitted 2007-04-03; First posted 2007-04-05 (Estimated); Last update posted 2007-09-17 (Estimated); Status verified 2007-09

CONDITIONS: Healthy
MeSH Terms: interventions — Fluvoxamine; Paroxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: AV650
Drug: Fluvoxamine
Drug: Paroxetine

SUMMARY:
The purpose of this study is to evaluate the effects that paroxetine and fluvoxamine have on the way the body distributes, breakdowns and eliminates AV650. In addition, information about any side effects that may occur will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18.5 to 29.9 kg/m2
* In good health, determined by no clinically significant findings from medical history, 12-lead ECG, and vital signs
* Clinical laboratory evaluations within the reference range for the test laboratory
* Negative test for selected drugs of abuse at Screening
* Negative HBsAg and HIV antibody screens
* Females of childbearing potential must be surgically sterile, post-menopausal for at least one year, or using and effective method of contraception; females of child bearing potential must have a negative serum pregnancy test at Screening and Day -1
* Males must be either sterile or agree to use an approved method of contraception
* Able to comprehend and willing to sign an Informed Consent Form

Exclusion Criteria:

* History or clinical manifestations of significant metabolic, hepatic, renal, hematological, pulmonary, cardiovascular, endocrine, gastrointestinal, urological, neurological, psychiatric disorders, or cancer
* History of inflammatory arthritis
* History of symptomatic hypotension
* History of severe physical injury, direct impact trauma, or neurological trauma within 6 months
* History of seizure disorders
* History of bipolar or major depressive disorder
* History of hypersensitivity or allergies to any drug compound
* Known intolerance to benzodiazepines
* Known intolerance to active and/or inactive ingredients in fluvoxamine or paroxetine
* History of stomach or intestinal surgery or resection, except that appendectomy, hernia repair, and/or cholecystectomy will be allowed
* History or presence of an abnormal ECG
* History of alcoholism, drug abuse, or drug addiction
* Use of any nicotine-containing or nicotine-replacement products within 6 months of Day -1
* Participation in any other investigational study drug trial within 90 days of Day -1
* Use of any prescription medications/products within 3 months of Day 1 unless deemed acceptable by the PI
* Received any vaccination or immunization within 1 month of Day -1
* Use of any over-the-counter, non-prescription preparations within 7 days of Day -1
* Use of alcohol-containing, grapefruit-containing, or caffeine-containing foods or beverages with 72 hours of Day -1
* Poor peripheral venous access
* Donation of blood within 3 months of Day -1 or of plasma within 2 weeks of Screening
* Receipt of blood products within 2 months of Day 1
* Female subjects who are pregnant or nursing
* Any acute or chronic condition that, in the opinion of the PI, would limit the subject's ability to complete and/or participate in this clinical study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-04; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of AV650

SECONDARY OUTCOMES:
Safety and tolerability of AV650
Genetic contribution, if any, to AV650 metabolism

CONTACTS AND LOCATIONS:
Locations (1):
- Covance Global Clinical Pharmacology Inc., San Diego, California, United States